CLINICAL TRIAL: NCT07258069
Title: Observational, Prospective, Multicenter Study On Histoacryl Used For Embolization Of Middle Meningeal Artery (MMA) In Chronic Subdural Hematoma (CSDH) (HARMONY)
Brief Title: Study On Histoacryl Used For Embolization Of Middle Meningeal Artery (MMA) In Chronic Subdural Hematoma (CSDH) (HARMONY)
Acronym: HARMONY
Status: Not yet recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-25118
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Subdural Hematoma; Subdural Hematoma, Chronic
MeSH Terms: conditions — Hematoma, Subdural; Hematoma, Subdural, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Histoacryl® — Histoacryl® is used by direct needle puncture, transcatheter approach, or transendoscopic approach in vascular embolization for the described purposes.

SUMMARY:
The aim of the study is to proof the effectiveness of Histoacryl® on preventing recurrence or progression of subdural hematoma after embolization of the middle meningeal artery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Confirmed diagnosis of chronic subdural hematoma (CSDH) or recurrent subdural hematoma (SDH)
* Completed documented informed consent
* Willingness and presumed capability to participate in follow-up visits for up to 6 months (180±30 days)

Exclusion Criteria:

* Extensive cerebral infarction, brain tumor, or space-occupying lesion requiring treatment
* Need craniotomy
* Any sign of anatomical variations that could make MMA embolization unsafe (e.g., prominent MMA-opthalmic artery anastomoses)
* Coagulation dysfunction with INR>1.8 and/or platelet count <80x109 /L
* Allergic reactions to essential medicines to do angiography
* Women who are pregnant, lactating, or who are of childbearing age and plan on becoming pregnant during the study
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A description of the population from which the groups or cohorts will be selected (for example, primary care clinic, community sample, residents of a certain town).
Sampling Method: Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence or progression of subdural hematoma | within 3 months
  Recurrence will be described as maximum thickness of SDH exceeding 10 mm, recurrence of symptoms or the patient requiring reoperation, meaning a second burr-hole drainage due to SDH.
  **Progression will be described as maximum thickness of SDH increasing over 3 mm compared to the baseline.

SECONDARY OUTCOMES:
Efficacy (1. Time) | V1, preoperatively (baseline visit)
  Time period from symptoms to embolization
Efficacy (2. Time) | V2, surgery (index procedure)
  Time period from burr-hole drainage to embolization
Efficacy (3. Time) | 6 months
  Time period from embolization to recurrence
Efficacy (4. Hematoma thickness) | at V4: 3 months and V5: 6 months compared to baseline
  Change in hematoma thickness
Efficacy (5. Change in midlind shift) | at V4: 3 months and V5: 6 months
  Change in midline shift compared to baseline
Efficacy (6. Cognitive assessment) | V1: preoperatively, V3: discharge, V4: 3 months and V5: 6 months
  Mini-Mental State Examination (MMSE) from 0 (severe cognitive impairment) to 30 (no cognitive impairment)
Quality of life, EQ-5D | V1: preoperatively, V3: discharge, V4: 3 months and V5: 6 months
  assessed by EQ-5D scale from 0 (worst health) to 100 (best health)

IPD SHARING:
Plan to Share IPD: No